CLINICAL TRIAL: NCT05756153
Title: A Phase Ib/II, Multi-Center, Open-Label Study to Evaluate the Safety/Tolerability, Pharmacokinetics, and Efficacy of GFH925 in Combination With Cetuximab in Previously Untreated Advanced NSCLC Harboring KRAS G12C Mutation
Brief Title: A Study of GFH925 in Combination With Cetuximab in Previously Untreated Advanced NSCLC Harboring KRAS G12C Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH925X0201
Record Dates: First submitted 2023-02-12; First posted 2023-03-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Advance Non-small Cell Lung Cancer
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GFH925+Cetuximab (Experimental)
  Interventions: Drug: GFH925; Drug: Cetuximab

INTERVENTIONS:
Drug: GFH925 — GFH925 tablets administered orally daily.
Drug: Cetuximab — Cetuximab administered intravenously Q2W.

SUMMARY:
This is a Phase Ib/II study. The objectives are to evaluate the safety/tolerability and efficacy of GFH925 in combination with Cetuximab in advanced KRAS G12C mutant NSCLC, to characterize pharmacokinetics (PK) of GFH925 in combination with Cetuximab in advanced KRAS G12C mutant NSCLC

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided informed consent form (ICF).
2. Males or females aged ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1.
4. Life expectancy > 3 months judged by the investigator.
5. Have histologically or cytologically confirmed advanced KRAS G12C-mutated NSCLC.
6. Have at least one measurable lesion per RECIST 1.1.
7. Have sufficient organ functions.
8. With toxicities left from prior anti-tumor therapy resolved to baseline or CTCAE Grade 1 (neurotoxicity or alopecia ≤ Grade 2).
9. Women of childbearing potential (WOCBP) and male patients with WOCBP partners must agree to use effective contraception method during the study specified period.

Exclusion Criteria:

1. With clinically significant cardiovascular diseases.
2. With active central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. With clinically significant gastrointestinal diseases.
4. With active infections.
5. With uncontrollable or symptomatic pleural effusion, ascites, or pericardial effusion.
6. With uncontrolled systemic diseases, such as hypertension or diabetes.
7. Prior treatment with an inhibitor specific to KRAS G12C.
8. Major surgery within 4 weeks prior to initiation of study treatment.
9. With known allergies to the study drugs or components.
10. Pregnant or lactating females, or female patients intend to become pregnant during participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Phase Ib: adverse events | 28 days
  defined as number of patients with treatment emergent AEs
Phase II: objective response rate | up to 1 year after last patient in
  defined as the percent of patients documented a PR/CR

CONTACTS AND LOCATIONS:
Locations (21):
- Greece (4):
  - University General Hospital "Attikon", Athens, Haidari
  - General Hospital of Athens "Alexandra", Athens
  - University General Hospital "Attikon", Athens
  - Bioclinic Thessaloniki, Thessaloniki
- Italy (8):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna, Emilia-Romagna
  - IRCCS Centro di Riferimento Oncologico, Aviano, Friuli Venezia Giulia
  - IOV - Istituto Oncologico Veneto IRCCS, Padova, Friuli Venezia Giulia
  - Istituto Nazionale Tumori Regina Elena IRCCS, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Candiolo Cancer Institute, FPO-IRCCS, Candiolo, Piedmont
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena, Tuscany
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma), Verona, Veneto
- Spain (9):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol,Servicio de Oncologia Medica, Badalona, Barcelona
  - Clinica Universidad de Navarra, Servicio de Oncologia, Pamplona, Navarre
  - Hospital Universitari Dexeus,Servicio de Oncologia Medica, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Clinica Mi Tres Torres, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Regional Universitario de Malaga,Oncology Dept, Málaga
  - Virgen del Rocio University Hospital, Seville
  - Instituto Valenciano de Oncologia IVO,Servicio de Oncologia Medica, Valencia